CLINICAL TRIAL: NCT00295308
Title: Clonidine for Relapse Prevention in Buprenorphine-Maintenance Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 999906407; 06-DA-N407
Record Dates: First submitted 2006-02-22; First posted 2006-02-23 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-09-17

CONDITIONS: Opioid-Related Disorders
Keywords: Opioid Dependence; Clonidine; Buprenorphine; Opioid Abstinence; Relapse
MeSH Terms: conditions — Opioid-Related Disorders; Recurrence | interventions — Clonidine

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Clonidine
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clonidine — clonidine up to 0.3 mg/day oral
  Arms: Arm 1
Drug: Placebo — oral capsules daily
  Arms: Arm 2

SUMMARY:
Background:

* Though the drug buprenorphine effectively treats dependence on opioids like heroin, some abstinent patients relapse to use during treatment. This relapse may be triggered by stress or stressful situations, and buprenorphine probably has no specific protective effect in these situations. Buprenorphine probably also has no specific effect on relapse to cocaine use.
* Research has shown that clonidine, a drug originally prescribed to treat high blood pressure and some symptoms of opioid withdrawal, can help block stress-induced relapse to heroin and cocaine seeking in rats. Researchers are interested in studying whether a combination of clonidine and buprenorphine may be more effective in preventing drug relapse than administering one of the medications alone.

Objectives:

- To determine whether clonidine, given to abstinent patients maintained on buprenorphine, is more effective than placebo in preventing relapse to heroin or cocaine use.

Eligibility:

- Individuals between 18 and 50 years of age who are current cocaine or heroin users seeking treatment.

Design:

* The study will last up to 36 weeks, with four phases of treatment and a follow-up evaluation. Three times a week, participants will be asked to report illicit drug use and provide urine and breath samples. Throughout the study, participants will receive individual counseling in weekly 40 60 minute sessions. Other samples and tests will be scheduled as required by the study researchers.
* Patients will be stabilized on daily buprenorphine over the first 14 days of the study.
* Weeks 1 8: Participants will receive vouchers for regular substance-free urine samples. Those who successfully complete this phase will continue to the next part of the study.
* Weeks 7 9: Participants will receive either clonidine or placebo along with the buprenorphine. The dose of clonidine will be stabilized during this time.
* Weeks 9 22: Participants will continue to receive either clonidine or placebo along with the buprenorphine. During this part of the study, participants will keep electronic diaries to record drug use or craving and to record data on mood, stress levels, and activity.
* Weeks 23 28: Participants will stop taking the clonidine or placebo, but will continue the buprenorphine treatment. Participants will continue to keep electronic diaries.
* Weeks 29 36: Participants will have the choice of transferring to a community clinic transfer or gradually reducing doses of buprenorphine to end the study.
* Participants will return for a follow-up visit and urine sample 6 months after the end of the study.

DETAILED DESCRIPTION:
Background. Though buprenorphine effectively treats opioid dependence, some abstinent patients relapse to maladaptive use of opioids during treatment. Relapse may be triggered by stress. Rodent studies have demonstrated that stress can induce relapse to heroin and cocaine use (Erb, et al., 1996; Shaham, et al., 1996; Shaham and Stewart, 1995). In a rodent model, stress-induced relapse to heroin and cocaine seeking is blocked by the alpha-2 adrenergic agonist clonidine. In this study, clonidine will be compared to placebo in preventing relapse to opioid abuse in opioid maintained patients who have achieved abstinence while on buprenorphine and contingency management.

Scientific goals. To determine whether clonidine, given to abstinent patients maintained on buprenorphine, prevents relapse to opioid use more effectively than placebo.

Participant population. 300 opioid-dependent outpatients (120 evaluable). Target enrollment will include 40 persent women and 60 percent minorities (mostly African-American).

Experimental design and methods. The study will be a randomized double-blind clinical trial. Two treatment groups will be studied (60/group), one receiving clonidine and the other receiving placebo. Assignment to treatment group will be randomized. All patients will receive buprenorphine daily (8 mg to 24 mg SL) and individual counseling weekly throughout 28 weeks of treatment. In order to establish abstinence prior to clonidine induction, after one week of stabilization on buprenorphine, they will receive contingent vouchers for opioid-negative urine specimens for 8 weeks (weeks 1-8). Patients who are abstinent from illicit opioids during weeks 5 and 6 will be randomized to receive clonidine (0.3 mg oral dose) or clonidine placebo from weeks 9 through 20. Participants who are not abstinent will be switched to methadone for four weeks (usual dose from 50 mg to 100 mg) followed by an eight week methadone taper. Assignment to clonidine or placebo will be double-blind. Weeks 21 and 22 will include a clonidine taper to avoid rebound hypertension. From weeks 23-28, participants will receive buprenorphine and counseling only, and then will be offered assistance to transfer to another program; those who do not transfer will undergo an 8-week buprenorphine taper. The primary outcome measures will be longest duration of opioid abstinence, time to relapse, and the proportion of opioid-negative urine specimens over time during the Intervention phase. In addition, fluctuations in drug use, drug craving, stress, and HIV-risk behaviors such as injection drug use will be assessed via ecological momentary assessment (EMA).

Benefits to participants and/or society. Participants will receive buprenorphine, drug counseling, and contingency-management therapy. The buprenorphine and voucher interventions are likely to reduce participants' use of opioids. Counseling will include reduction of HIV risk behaviors.

Risks to participants. Participants may experience side effects from clonidine, buprenorphine, or methadone and discomfort during withdrawal from each drug. In particular, discontinuation of clonidine may cause rebound hypertension. The EMA component of the study may generate some assessment burden.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age between 18 and 60
  2. Evidence of physical dependence on opioids (self-report, urine screen, physical exam)
  3. Seeking treatment for opioid dependence
  4. Able to attend treatment clinic 7 days/week

EXCLUSION CRITERIA:

General-

1. Poor venous access
2. Urologic conditions that would inhibit urine collection
3. Pregnancy or breastfeeding
4. Failure to agree to use a medically effective form of contraception while in the study (in women who are sexually active with a male partner and able to get pregnant). Acceptable forms of contraception for this study include: hormonal contraceptives (birth control pills, injectable hormones, vaginal ring hormones), surgical sterility (tubal ligation or hysterectomy); IUD; Diaphragm with spermicide; Condom with spermicide
5. Current physical dependence on alcohol or sedative-hypnotics, e.g. benzodiazepines

Psychiatric-

1. Cognitive impairment severe enough to preclude informed consent or valid responses on questionnaires (Shipley Institute of Living scale estimated full-scale IQ less than 80)
2. History of schizophrenia or any other DSM-IV psychotic disorder
3. History of bipolar disorder
4. Current Major Depressive Disorder

Medical-

1. Any active or untreated medical illness that in the view of the investigators would compromise participation in research
2. Allergy or intolerance to either buprenorphine or clonidine
3. Cerebrovascular disease
4. Conduction disturbances (e.g., second-degree heart block, third-degree heart block, atrial fibrillation, ventricular tachycardia) or arrhythmias
5. Myocardial infarction, or documented coronary artery disease
6. Congestive heart failure
7. Chronic renal failure, as estimated by Cr > 2.0
8. CD4 < 200 or evidence of severely compromised immune system /AIDS
9. Marked, sustained bradycardia (HR < 45 bpm) on three separate occasions
10. Marked, sustained low blood pressure (SBP <95 or DBP < 40 mm Hg) over three separate readings
11. Marked, sustained high blood pressure (SBP >160 mm Hg, DBP >100 mm Hg) over several readings, without being on antihypertensive medications.
12. ECG changes suggestive of acute ischemia, clinical important arrhythmia, left bundle branch block, or other changes that concerns the MRP will exclude the participant. If accompanied by cardiovascular complaints such as chest pain or syncope, less specific ECG findings will also exclude the patient. When in doubt, the ECG will be sent to cardiology on a prn basis for a manual reading.
13. Orthostatic hypotension (upon standing for 3 minutes, there is a 20 mm Hg decrease in systolic blood pressure or a 10 mmHg decrease in diastolic blood pressure accompanied by an increase by 20 bpm in heart rate) on two separate readings.

Taking contraindicated medications-

1. Beta blockers
2. Tricyclic antidepressants
3. Antipsychotics
4. Mah huang
5. Yohimbe
6. Ephedra
7. Sildenafil citrate (Viagra). Sildenafil citrate doses > 25mg should not be taken within 4 hours of taking an alpha blocker or it can produce significant and symptomatic hypotension (Pfizer). Of note, Viagra, like buprenorphine, is metabolized by cytochrome P450 3A4. Ingestion of buprenorphine could potentate the effects of sildenafil citrate which could extent the period of safety to > 4 hrs from when an alpha blocker could be taken after Viagra ingestion.

Family history of sudden cardiac death at age < 50

Lab Test and Lab Values:

WBC* < 1,500 > 13,000 #/CUMM

HCT < 33 > 49 Percent

Platelets < 100 > 500 K/CUMM

Sodium < 132 > 149 MEQ/L

Potassium < 3.5 > 5.2 MEQ/L

Calcium < 8.4 > 10.5 MG/DL

Magnesium < 1.3 > 3 MG/DL

<TAB>

BUN > 35 MG/DL

Cr<TAB> > 2.0 MG/DL

<TAB>

Alk Phos<TAB> > 200 U/L

AST<TAB> > 200 U/L

ALT<TAB> > 200 U/L

GGT<TAB> > 400 U/L

Albumin<TAB> < 3 GM/DL

Total bilirubin > 2.0 MG/DL

Direct bilirubin > 0.4 MG/DL

TSH<TAB> < 0.27 > 4.2 UIU/ML

<TAB>

*Leukocytosis will prompt further investigation before clearance.<TAB>

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 208 (Actual)
Dates: Start 2005-11-08; Study Completion 2014-07-30 (Actual)

PRIMARY OUTCOMES:
Opiate-negative urine screens | 38 weeks

SECONDARY OUTCOMES:
HIV risk behaviors | 38 weeks
Craving | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kenzie Preston, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Kowalczyk WJ, Moran LM, Bertz JW, Phillips KA, Ghitza UE, Vahabzadeh M, Lin JL, Epstein DH, Preston KL. Using ecological momentary assessment to examine the relationship between craving and affect with opioid use in a clinical trial of clonidine as an adjunct medication to buprenorphine treatment. Am J Drug Alcohol Abuse. 2018;44(5):502-511. doi: 10.1080/00952990.2018.1454933. Epub 2018 Apr 10. PMID 29634425
- [Derived] Kowalczyk WJ, Phillips KA, Jobes ML, Kennedy AP, Ghitza UE, Agage DA, Schmittner JP, Epstein DH, Preston KL. Clonidine Maintenance Prolongs Opioid Abstinence and Decouples Stress From Craving in Daily Life: A Randomized Controlled Trial With Ecological Momentary Assessment. Am J Psychiatry. 2015 Aug 1;172(8):760-7. doi: 10.1176/appi.ajp.2014.14081014. Epub 2015 Mar 17. PMID 25783757